CLINICAL TRIAL: NCT03804892
Title: Can Brisk Walking Combined With Ingestion of a Lipid-lowering Drug Improve Fat Metabolism in Muscle?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Diabetes UK (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Royal Liverpool University Hospital (Other Government)
Responsible Party: Principal Investigator, Jennifer Barrett, PhD researcher in Exercise Metabolism, Liverpool John Moores University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 249734
Record Dates: First submitted 2019-01-07; First posted 2019-01-15 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Body Composition; Glucose Tolerance Test; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This study involves 2 trials. Each trial will involve walking for 45 minutes on a treadmill, with muscle biopsies obtained from the thigh before (basal), immediately following (post-exercise) and 3 h post-exercise. Each trial will be identical, except that participants will ingest either Acipimox or a placebo in a double-blind design. Muscle biopsies will be used to examine differences in muscle fat between the two trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acipimox ingestion (Experimental): Participants will undergo pre assessment testing of a body composition (DEXA), a maximal aerobic fitness test, and an oral glucose tolerance test. Following this, participants will ingest 250 mg of Acipimox, before undertaking 45 minutes walking on a treadmill. A muscle biopsy will be taken pre, immediately post and 3 hours post the walking trial. Blood samples will be taken at regular intervals throughout.
  Interventions: Diagnostic Test: Body Composition; Diagnostic Test: Maximal aerobic fitness test; Diagnostic Test: Oral glucose tolerance test; Other: Muscle biopsy; Other: Blood samples
- No drug (Other): Participants will undergo pre assessment testing of a body composition (DEXA), a maximal aerobic fitness test, and an oral glucose tolerance test.Participants will then undergo a 45 minute walk on a treadmill with no Acipimox ingestion. A muscle biopsy will be taken pre, immediately post and 3 hours post the walking trial. Blood samples will be taken at regular intervals throughout.
  Interventions: Diagnostic Test: Body Composition; Diagnostic Test: Maximal aerobic fitness test; Diagnostic Test: Oral glucose tolerance test; Other: Muscle biopsy; Other: Blood samples

INTERVENTIONS:
Diagnostic Test: Body Composition — Participants undergo a 5 minute body scan to determine their body composition.
Diagnostic Test: Maximal aerobic fitness test — Participants will complete a walking fitness text until exhaustion to determine maximal aerobic capacity.
Diagnostic Test: Oral glucose tolerance test — Participants will undergo an OGTT to determine insulin sensitivity.
Other: Muscle biopsy — Participants will give a small muscle sample pre-, immediately post and 3 hours post- the exercise trial to be assessed for lipid metabolites.
Other: Blood samples — Participants will give 16 blood samples, to be assessed for fatty acids in the blood.

SUMMARY:
Briefly, participants will be assessed for their eligibility for the study using an oral glucose tolerance test, which involves drinking a sugary drink followed by a series of small blood samples. If eligible, participants will be asked to take part in a fitness test and then two trials which will involve walking on a treadmill at a steady pace. Before and after the exercise a small piece of muscle will be taken from their thigh under local anaesthesia, as well as several small blood samples. Muscle muscle samples will be assessed for lipid metabolites.

DETAILED DESCRIPTION:
The accumulation of fat in skeletal muscle is linked with insulin resistance in obesity and T2D. However, fat also accumulates in the muscle of lean, healthy people, but they remain insulin sensitive. This is because healthy people are able to burn this fat to generate energy during exercise. However, overweight/obese inactive people can't use muscle fat during exercise in the same manner, which is related to the high blood lipid concentrations that are observed in these individuals. Acipimox is a lipid-lowering agent that specifically reduces the breakdown of fat in adipose tissue and has been shown improve the blood lipid profile of obese individuals and T2D patients, at least in the short-term (1-2 weeks). Previous research has shown that the combination of Acipimox with exercise restores the ability of obese people to burn fat during moderate-intensity cycling exercise. It is now important to test whether Acipimox also increases the ability to burn muscle fat during low-intensity walking in people with prediabetes. If it does, then the next step will be to test whether the combination of Acipimox and walking can lead to improved insulin sensitivity and reduced T2D risk over a longer intervention programme. Twelve people with pre-diabetes will be recruited to undertake two experimental trials in a randomised order. Each trial will involve walking for 45 minutes on a treadmill, with muscle biopsies obtained from the thigh before (basal), immediately following (post-exercise) and 3 h post-exercise. Each trial will be identical, except that participants will ingest either Acipimox or a placebo in a double-blind design. Muscle biopsies will be used to examine differences in muscle fat between the two trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25-55 years
* Overweight or obese (BMI >28 kg.m-2)
* Have prediabetes
* Not currently using any anti-diabetes medication
* Physically inactive (performing less than two 30 min structured exercise sessions per week for the last year)
* Not pregnant (or intending to get pregnant during the study) or currently breast feeding
* Pre-menopausal
* Not currently involved in a weight loss programme or using weight loss medication

Exclusion Criteria:

* Involved in regular exercise (engaged in more than 2 sessions of structured exercise of >30 min per week)
* Currently using anti-diabetes medication (e.g. insulin, metformin)
* Currently using niacin/vitamin B3 supplements
* Pregnant or breast feeding
* Currently engaged in active weight loss programmes or using weight loss medication
* Diagnosed with chronic kidney disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Plasma fatty acids levels | A change in the amount of fatty acids in the blood from baseline, to every 15 minute interval from the ingestion of acipimox up until 2 hours 45 minutes. From this point, samples will be every 30 minutes until 3 hours 45 minutes terminates the trial.
  Blood samples will be assessed for the amount of fatty acids in the blood.
Skeletal muscle Diacylglycerol (DAG) levels | A change from baseline DAGs to DAGS immediately post and 3 hours post exercise trial.
  Muscle biopsies will be assessed for lipid metabolites using liquid chromatography-mass spectrometry.
Plasma Glycerol levels | A change in the amount of fatty acids in the blood from baseline, to every 15 minute interval from the ingestion of acipimox up until 2 hours 45 minutes. From this point, samples will be every 30 minutes until 3 hours 45 minutes terminates the trial.
  Blood samples will be assessed for the amount of glycerol in the blood throughout the exercise trial.
IMTG utilisation during exercise | A change in amount of IMTG within the muscle from baseline, to immediately post and 3 hours post the exercise intervention.
  Muscle samples will be analysed using confocal immunofluorescence microscopy for the amount of IMTG within the samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Barrett, PhD, Principal Investigator — Liverpool John Moores University, L3 3AF
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No